CLINICAL TRIAL: NCT03116763
Title: The iPeer2Peer Program for Adolescents With Juvenile Idiopathic Arthritis: A Randomized Controlled Trial
Brief Title: The iPeer2Peer Program for Adolescents With Juvenile Idiopathic Arthritis
Acronym: iPeer2Peer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Provincial Health Services Authority British Columbia (Other); IWK Health Centre (Other); Children's Hospital of Eastern Ontario (Other)
Responsible Party: Principal Investigator, Jennifer Stinson, Senior Scientist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1000054878
Record Dates: First submitted 2017-03-31; First posted 2017-04-17 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Juvenile Idiopathic Arthritis
MeSH Terms: conditions — Arthritis, Juvenile

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iPeer2Peer Mentorship (Experimental): In addition to standard care, youth in the experimental group will receive the iPeer2Peer program, a peer mentorship program that will provide modeling and reinforcement of self-management by pre-screened and trained peer mentors (young adults with JIA aged 18-22 years who have learned to function successfully with their disease). Mentors will encourage participants to develop and engage in self-management skills and provide social support.
  Interventions: Behavioral: iPeer2Peer Mentorship
- Control Group (Active Comparator): The control group will receive standard care but without the iPeer2Peer program.
  Interventions: Other: Active Comparator: Control Group

INTERVENTIONS:
Behavioral: iPeer2Peer Mentorship — 10 sessions of 20-30 minute Skype calls conducted over 5-12 weeks.
  Arms: iPeer2Peer Mentorship
Other: Active Comparator: Control Group — The control group will receive standard care but without the iPeer2Peer program.
  Arms: Control Group

SUMMARY:
The iPeer2Peer program matches teens with arthritis to an older mentor who has learned to manage their arthritis well and can support them emotionally and socially. This study will compare two groups of teens: those who are in the iPeer2Peer Program and those in the control group (no mentor).

DETAILED DESCRIPTION:
Arthritis is a common childhood illness that makes everyday activities hard for young people. It is a long-lasting illness that can make you feel pain, tired and emotionally upset. This can make it hard for children and teens to see friends and do the activities that they like. The goal of this project is to find out if the newly developed peer mentoring program called iPeer2Peer helps teens with arthritis take better care of their illness and feel more connected to other people with arthritis. The iPeer2Peer program matches teens with arthritis to an older mentor who has learned to manage their arthritis well and can support them emotionally and socially. This study will compare two groups of teens: those who are in the iPeer2Peer Program and those in the control group (no mentor).

ELIGIBILITY:
Inclusion Criteria:

* males and females 12-18 years old
* rheumatologist-diagnosed JIA according to ILAR criteria
* able to speak and read English
* access to a computer, smartphone or tablet capable of using free Skype software (note: participants who do not have adequate Internet access will be provided with portable Internet sticks)
* willing and able to complete online measures.

Exclusion Criteria:

* significant cognitive impairments
* major co-morbid illnesses (medical or psychiatric conditions) likely to influence HRQL assessment
* participating in other peer support or self-management interventions.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 164 (Actual)
Dates: Start 2017-03-28 (Actual); Primary Completion 2023-04-16 (Actual); Study Completion 2023-04-16 (Actual)

PRIMARY OUTCOMES:
TRANSITION-Q (measuring change) | Baseline; Immediately following interview (approximately 12 weeks after baseline); 6-months post
  14-item measure of self-management skills that is both reliable (internally consistent, test-retest) and valid (face, construct and content validity)

SECONDARY OUTCOMES:
PedsQL Arthritis Module (measuring change) | Baseline; Immediately following interview (approximately 12 weeks after baseline); 6-months post
  Health-related quality of life
PROMIS Pain Interference (measuring change) | Baseline; Immediately following interview (approximately 12 weeks after baseline); 6-months post
  Pain
Screen for Child Anxiety Related Disorders (measuring change) | Baseline; Immediately following interview (approximately 12 weeks after baseline); 6-months post
  Emotional distress
Center for Epidemiologic Studies Depression Scale Revised (measuring change) | Baseline; Immediately following interview (approximately 12 weeks after baseline); 6-months post
  Emotional distress
Medical Issues, Exercise, Pain and Social Support Questionnaire (measuring change) | Baseline; Immediately following interview (approximately 12 weeks after baseline); 6-months post
  Disease knowledge
Children's Arthritis Self-Efficacy (measuring change) | Baseline; Immediately following interview (approximately 12 weeks after baseline); 6-months post
  Self-efficacy
PROMIS Pediatric Peer Relationship Scale (measuring change) | Baseline; Immediately following interview (approximately 12 weeks after baseline); 6-months post
  Perceived social support
AQoL-6D, interview (measuring change) | Baseline; Immediately following interview (approximately 12 weeks after baseline); 6-months post
  Cost utility analysis
Health service use and costs (measuring change) | Baseline; Immediately following interview (approximately 12 weeks after baseline); 6-months post
  Cost utility analysis
Mentor Behavior Scale (measuring change) | Post-Intervention (approximately following 12 weeks of calls)
  Mentor quality
PROMIS Adult Profile (measuring change) | At beginning of study and at end of study (approximately 3 years later)
  For mentors only: mentor physical and emotional symptoms
PROMIS Satisfaction with Social Roles and Activities (measuring change) | At beginning of study and at end of study (approximately 3 years later)
  For mentors only: perceived social role satisfaction
Chronic Disease Self-Efficacy Scale (measuring change) | At beginning of study and at end of study (approximately 3 years later)
  For mentors only: self-efficacy
Mentor interaction form | Following completion of each mentee's calls (approximately following 12 weeks of calls)
  Record of interactions with mentees

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer N Stinson, CPNP, PhD, Principal Investigator — The Hospital for Sick Children
Locations (6):
- Canada (6):
  - Alberta Children's Hospital, Calgary, Alberta
  - BC Children's Hospital, Vancouver, British Columbia
  - The IWK Health Centre, Halifax, Nova Scotia
  - Children's Hospital - London Health Sciences, London, Ontario
  - Children's Hospital of Eastern Ontario (CHEO), Ottawa, Ontario
  - The Hospital for Sick Children, Toronto, Ontario

REFERENCES:
- [Derived] Nishat F, Kelenc L, Berard R, Duffy C, Feldman B, Forgeron P, Huber AM, Luca N, Schmeling H, Spiegel L, Tucker L, Watanabe-Duffy K, Killackey T, Lalloo C, Wiles B, Nair A, Olaizola S, McDermott B, Tavangar F, Kohut SA, Stinson JN. Assessing the impact of the iPeer2Peer program for adolescents with juvenile idiopathic arthritis: a mixed-methods randomized controlled trial. Pediatr Rheumatol Online J. 2024 Dec 27;22(1):109. doi: 10.1186/s12969-024-01052-5. PMID 39731098